CLINICAL TRIAL: NCT04381013
Title: Emergency Ventilator Splitting Between Two or More Patients Using a Single Ventilator to Address Critical Ventilator Shortages During a Pandemic
Brief Title: Emergency Ventilator Splitting Between Two or More Patients (COVID-19)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Different approach to be taken for the device.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 57573
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Phase 1: Routine surgery (Experimental): As part of routine cardio-thoracic surgery, endotracheal tubes split from ventilator delivering oxygen independently to each lung for up to 1 minute.
  Interventions: Device: Emergency Ventilator Splitter
- Phase 2: ECHO treatment (Experimental): During care with Extracorporeal Membrane Oxygenation (ECMO) for non-SARS-CoV-2, endotracheal tubes split from ventilator delivering oxygen independently to each lung for up to 24 hours.
  Interventions: Device: Emergency Ventilator Splitter
- Phase 3: COVID-19 treatment (Experimental): Endotracheal tubes split from ventilator delivering oxygen independently to two patients with COVID-19 disease for up to 1 hour.
  Interventions: Device: Emergency Ventilator Splitter

INTERVENTIONS:
Device: Emergency Ventilator Splitter — Device to enable oxygen delivery to two patients independently from a single ventilator.

SUMMARY:
The purpose of this study is to develop a safe, easily scalable, and simple method to split a single ventilator for use amongst two or more patients, thus serving as a capacity bridge to save patient lives until manufacturers can produce enough ventilators.

ELIGIBILITY:
Inclusion Criteria:

* Phase I

  * Undergoing routine thoracic surgery which will include the use of a dual lumen endotracheal tube at Stanford.
* Phase II

  * Able to give consent
  * On venovenous extracorporeal membrane oxygenation for reason other than COVID-19
* Phase III

  * Able to give consent
  * Infected with COVID-19 and will likely require mechanical ventilation.

Exclusion Criteria:

* Phase I

  * Significant cardiac comorbidities
  * Liver disease
* Phase II

  * Significant cardiac comorbidities
  * Pre or Post-transplant patient
  * Infection with COVID-19
* Phase III

  * Co-infection with disease aside from COVID-19
  * Severely ill requiring high ventilator requirements and not stable for ventilator splitting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Completion of 1-minute test | Up to 1 minute
  This outcome will measure whether the device will function for respiratory support for 1 minute (yes or no; phase 1 only)
Completion of 24-hour test | Up to 1 minute
  This outcome will measure whether the device will function for respiratory support for 24 hours (yes or no; phase 2 only)
Completion of 24-hour test | Up to 1 hour
  This outcome will measure whether the device will function for respiratory support for 1 hour (yes or no; phase 3 only)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Woo, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.